CLINICAL TRIAL: NCT03520803
Title: A Prospective Randomized Study of an Enhanced Recovery After Surgery Pathway in Patients Undergoing Laparoscopic Sleeve Gastrectomy
Brief Title: Enhanced Recovery After Surgery in Laparoscopic Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HHC-2017-0146
Record Dates: First submitted 2018-04-05; First posted 2018-05-11 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Obesity
Keywords: obesity; bariatric surgery; enhanced recovery after surgery; sleeve gastrectomy; gastric bypass
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): ERAS protocol
  Interventions: Other: Enhanced recovery after surgery protocol
- Control (No Intervention): Standard of care

INTERVENTIONS:
Other: Enhanced recovery after surgery protocol — Experimental enhanced recovery protocol for pre-surgery and post surgery
  Other Names: ERAS
  Arms: Experimental

SUMMARY:
While laparoscopic sleeve gastrectomy (LSG) has become the most commonly performed bariatric surgery procedure in the US and worldwide, it is associated with significant postoperative nausea and vomiting (PONV), which can lead to patient readmission for rehydration and symptom control. Enhanced recovery after surgery (ERAS) is an approach that aligns the practice of anesthesia with the care given by the surgical team before, during, and after surgery. A number of prospective series, retrospective analyses and one randomized clinical trial of ERAS use in bariatric patients support the idea that ERAS in this population is feasible, effective and safe and that it is associated with shorter lengths of stay, fewer readmissions and decreased costs. In this protocol, the investigators will conduct a prospective, randomized control study using a structured and integrative perioperative plan (ERAS; n = 64) vs. current standard of care (SOC; n = 64) for patients undergoing LSG at Hartford Hospital. The investigators are guided by the idea that an enhanced recovery protocol can potentially serve to enhance the early patient experience and set the stage for a more rapid transition out of the recovery phase and into the weight loss phase of the patient's care. The investigators will incorporate a postoperative multidrug strategy targeting multiple receptors to decrease PONV and pain, similar to ERAS Society recommendations for bariatric patients.

Specific Aims and Hypotheses The central hypothesis is that the introduction of an ERAS pathway in patients undergoing LSG is feasible and will lead to better clinical outcomes.

Aim 1. To evaluate the effect that introducing an ERAS pathway will have on the use of narcotic medication for the management of postoperative pain, PONV, readiness for discharge, and overall length of stay in patients undergoing LSG.

Aim 2. To evaluate the safety of the ERAS protocol by measuring inpatient and 30-day adverse events, emergency department (ED) visits, outpatient hydration, readmission rates and delirium.

Participants will be recruited through fliers posted at Surgical Weight Loss Center locations (Glastonbury, Enfield, Hartford, Farmington, Manchester and South Windsor).

ELIGIBILITY:
Inclusion Criteria:

• Patients scheduled to have laparoscopic sleeve gastrectomy at our surgical weight loss center

Exclusion Criteria:

* Participants whose primary language is not English;
* Patients who are wheel chair-bound and those who are on dialysis with end stage renal disease;
* Patients who have known allergic reactions to any of the ERAS protocol medications, which upon review by the clinical team are deemed clinically significant;
* Patients with a history of cardiac events or a prolonged QTc interval on preoperative EKG which could in the opinion of the investigators increase their risk for prolonged QTc interval when certain ERAS medications are given in combination;
* Patients who have chronic kidney disease (contraindication to use NSAIDs) or are currently taking narcotic pain medications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2019-01-26 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Rate of post-operative administration of narcotics or rescue anti-nausea medications | 1 week
  Including dilaudid, zofran, haldol, phenergan, ketorolac, remeron
Readiness for discharge | 1 day
  Readiness for discharge score: Taking 5 factors into account. Scores can range from 0 to 5 with a higher score representing higher readiness for discharge.
Hospital length of stay | 1 week
  Total length of stay in the hospital in days

SECONDARY OUTCOMES:
Adverse events | Measured continuously throughout hospital stay up to 30 days post discharge
  Total number of inpatient and 30 - day adverse events
Delirium | 1 week
  Delirium as measured using the Confusion Assessment Method

OTHER OUTCOMES:
BMI | Baseline
  Body mass index
Pain | 1 week
  Measured using the Pain Numeric Rating Scale. Patients are asked to rate their current pain with a low score representing less pain and a high score representing more pain Scores range from 0 - 10, as follows 2= mild pain, does not limit activities; 4= moderate pain, can do most activities with rest; 6= unable to do some activities because of pain; 8= severe pain, unable to do most activities because of pain; 10 = excruciating, unable to do any activities because of pain
Post-operative nausea and vomiting | 1 week
  Measured using the Postoperative Nausea and Vomiting Impact Scale. Scores range from 0 - 6, >/= 5 indicates clinically important post-operative nausea/vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Pavlos K Papasavas, MD, Principal Investigator — Hartford Hospital
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided